## หนังสือแสดงเจตนายินยอมเข้าร่วมการวิจัย

(Consent Form)

| | | วันที่เดือน | พ.ศ | |
|---------------------|---------|--------------|------|---|
| ข้าพเจ้า | | | อายุ | า |
| อาศัยอยู่บ้านเลขที่ | ถนน | แขวง/ตำบล | | |
| เขต/อำเภอ | จังหวัด | รหัสไปรษณีย์ | Í | |
| โทรศัพท์ | | | | |

ขอแสดงเจตนายินยอมเข้าร่วมโครงการวิจัย เรื่อง การศึกษาผลของยา Zolpidem ต่อการปรับตัวต่อเครื่องอัดอากาศแรงดันบวกในผู้ป่วยโรคหยุดหายใจขณะหลับจากการอุดกั้น: การทดลองแบบสุ่มไขว้และมีกลุ่มควบคุม

โดยข้าพเจ้าได้รับทราบรายละเอียดเกี่ยวกับที่มาและจุดมุ่งหมายในการทำวิจัย รายละเอียด ขั้นตอนต่าง ๆ ที่จะต้องปฏิบัติหรือได้รับการปฏิบัติ ประโยชน์ที่คาดว่าจะได้รับของการวิจัย และความ เสี่ยงที่อาจจะเกิดขึ้นจากการเข้าร่วมการวิจัย รวมทั้งแนวทางป้องกันและแก้ไขหากเกิดอันตรายขึ้น ค่าตอบแทนที่จะได้รับ 200 บาท เมื่อมาติดตามอาการครั้งที่ 1 และ 200 บาท เมื่อมาติดตามอาการครั้งที่ 2

โดยได้อ่านข้อความที่มีรายละเอียดอยู่ในเอกสารชี้แจงผู้เข้าร่วมการวิจัยโดยตลอด อีกทั้งยังได้รับ คำอธิบายและตอบข้อสงสัยจากหัวหน้าโครงการวิจัยเป็นที่เรียบร้อยแล้ว

ข้าพเจ้าจึงสมัครใจเข้าร่วมในโครงการวิจัยนี้

หากข้าพเจ้ามีข้อข้องใจเกี่ยวกับขั้นตอนของการวิจัย หรือหากเกิดผลข้างเคียงที่ไม่พึงประสงค์ จากการวิจัยขึ้นกับข้าพเจ้า ข้าพเจ้าจะสามารถติดต่อกับ แพทย์หญิงปิยากร พิศาลนรเดช ภาควิชาโสต นาสิก ลาริงซ์วิทยา คณะแพทยศาสตร์ ศิริราชพยาบาล มหาวิทยาลัยมหิดล 0818863677

หากข้าพเจ้าได้รับการปฏิบัติไม่ตรงตามที่ระบุไว้ในเอกสารชี้แจงผู้เข้าร่วมการวิจัย ต้องการ ปรึกษาปัญหา ข้อกังวล มีคำถามหรือต้องการข้อมูลเพิ่มเติมเกี่ยวกับการวิจัย ข้าพเจ้าสามารถติดต่อกับ ประธานคณะกรรมการจริยธรรมการวิจัยในคนได้ที่ สำนักงานคณะกรรมการจริยธรรมการวิจัยในคน อาคารเฉลิมพระเกียรติ ๘๐ พรรษา ๕ ธันวาคม ๒๕๕๐ ชั้น 2 โทร.0 2419 2667-72 โทรสาร 0 2411 0162

ข้าพเจ้าได้ทราบถึงสิทธิ์ที่ข้าพเจ้าจะได้รับข้อมูลเพิ่มเติมทั้งทางด้านประโยชน์และโทษจากการ เข้าร่วมการวิจัย และสามารถถอนตัวหรืองดเข้าร่วมการวิจัยได้ทุกเมื่อโดยไม่ต้องแจ้งล่วงหน้าหรือระบุ เหตุผล โดยจะไม่มีผลกระทบต่อการบริการและการรักษาพยาบาลที่ข้าพเจ้าจะได้รับต่อไปในอนาคต และยินยอมให้ผู้วิจัยใช้ข้อมูลส่วนตัวของข้าพเจ้าที่ได้รับจากการวิจัย แต่จะไม่เผยแพร่ต่อสาธารณะเป็น รายบุคคล โดยจะนำเสนอเป็นข้อมูลโดยรวมจากการวิจัยเท่านั้น

ข้าพเจ้าได้เข้าใจข้อความในเอกสารชี้แจงผู้เข้าร่วมการวิจัย และหนังสือแสดงเจตนายินยอมนี้ โดยตลอดแล้ว จึงลงลายมือชื่อไว้เป็นหลักฐาน ทั้งนี้ ข้าพเจ้าได้รับสำเนาหนังสือแสดงเจตนายินยอมเข้า ร่วมในการวิจัยไว้แล้ว 1 ฉบับ

| ลงชื่อ | ผู้ร่วมวิจัย/อาสาสมัครหรือผู้แทนโดยชอบธรรม/วันที่ |
|---|---|
| ( | ) |
| ลงชื่อ | ผู้ให้ข้อมูลและขอความยินยอม/หัวหน้าโครงการวิจัย/วันที่<br>) |
| ในกรณีผู้ร่วมวิจัย/อาสาสมัคร อ่านเ | หนังสือไม่ออก มีพยานซึ่งไม่มีส่วนได้เสียอยู่ด้วยตลอดระยะเวลาที่มีการให้ |
| ข้อมูลและผู้ร่วมวิจัย/อาสาสมัครหรือ | ผู้แทนโดยชอบธรรมให้ความยินยอมเข้าร่วมการวิจัย พยานขอยืนยันว่าข้อมูล |
| ในหนังสือแสดงเจตนายินยอมหรือ | ข้อมูลที่ได้รับและเอกสารอื่นได้รับการอธิบายอย่างถูกต้อง และผู้ร่วมวิจัย/ |
| อาสาสมัครหรือผู้แทนโดยชอบธรรมเ | แสดงว่าเข้าใจรายละเอียดต่างๆ พร้อมทั้งให้ความยินยอมโดยสมัครใจ จึงได้ |
| ลงลายมือชื่อไว้เป็นพยาน | |
| ลงชื่อ | พยาน/วันที่ |
| / | <b>\</b> |